CLINICAL TRIAL: NCT05480475
Title: A Single-center, Open-label, Three-period, Fixed-sequence Design Study to Investigate the Effect of Daridorexant on the Pharmacokinetics of Dabigatran and Rosuvastatin in Healthy Male Subjects
Brief Title: A Study to Examine the Effect of Daridorexant on the Way the Body Absorbs, Distributes, and Gets Rid of Dabigatran and Rosuvastatin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ID-078-125
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — Dabigatran; Rosuvastatin Calcium; daridorexant

STUDY DESIGN:
Intervention Model Description: Three-period, fixed-sequence design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Study treatment (Period 1, 2, and 3) (Experimental): Period 1: Treatment A1 - dabigatran etexilate; Treatment A2 - rosuvastatin Period 2: Treatment B - daridorexant Period 3: Treatment C1 - dabigatran etexilate and daridorexant; Treatment C2 - rosuvastatin and daridorexant
  Interventions: Drug: Dabigatran etexilate; Drug: Rosuvastatin; Drug: Daridorexant

INTERVENTIONS:
Drug: Dabigatran etexilate — On Day 1 (Treatment A1) and on Day 9 (Treatment C1) a single oral dose of 75 mg dabigatran etexilate will be administered under fasted conditions.
Drug: Rosuvastatin — On Day 3 (Treatment A2) and on Day 11 (Treatment C2) a single oral dose of 10 mg rosuvastatin will be administered under fasted conditions.
Drug: Daridorexant — On Day 7 and Day 8 (Treatment B), on Day 9 and Day 10 (Treatment C1), and on Day 11 through 14 (Treatment C2) subjects will receive 50 mg daridorexant o.d. under fasted conditions.

SUMMARY:
A study to examine the effect of daridorexant on the way the body absorbs, distributes, and gets rid of dabigatran and rosuvastatin in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
2. Healthy male subject aged between 18 and 45 years (inclusive) at Screening.

Exclusion Criteria:

1. Known hypersensitivity to daridorexant, rosuvastatin, and/or dabigatran etexilate, or treatments of the same class, or any of its/their excipients.
2. Any history of hemorrhagic disease, whether or not hereditary.
3. Any history of complications with bleeding after surgery or tooth extractions and/or frequent nasal, hemorrhoidal, or gingival bleeding.
4. Activated partial thromboplastin time (aPTT) and/or thrombin time (TT) < 0.8 or > 1.2 at Screening.
5. Clinically relevant findings on the physical examination at Screening.
6. Clinically relevant findings on 12-lead ECG, recorded after 5 min in a supine position at Screening.
7. Clinically relevant findings in clinical laboratory tests (hematology, coagulation, clinical chemistry, and urinalysis) at Screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-03 (Actual); Primary Completion 2022-09-17 (Actual); Study Completion 2022-09-17 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of dabigatran | Blood samples for pharmacokinetic analyses will be taken at various time points from Day 1 to 7 and Day 9 to 15 (total duration: 14 days).
Cmax of rosuvastatin | Blood samples for pharmacokinetic analyses will be taken at various time points from Day 1 to 7 and Day 9 to 15 (total duration: 14 days).

OTHER OUTCOMES:
Time to reach Cmax (tmax) of dabigatran | Blood samples for pharmacokinetic analyses will be taken at various time points from Day 1 to 7 and Day 9 to 15 (total duration: 14 days).
Tmax of rosuvastatin | Blood samples for pharmacokinetic analyses will be taken at various time points from Day 1 to 7 and Day 9 to 15 (total duration: 14 days).
Area under the plasma concentration-time curve from zero to infinity (AUC0-inf) of dabigatran | Blood samples for pharmacokinetic analyses will be taken at various time points from Day 1 to 7 and Day 9 to 15 (total duration: 14 days).
AUC0-inf of rosuvastatin | Blood samples for pharmacokinetic analyses will be taken at various time points from Day 1 to 7 and Day 9 to 15 (total duration: 14 days).
Terminal half-life (t½) of dabigatran | Blood samples for pharmacokinetic analyses will be taken at various time points from Day 1 to 7 and Day 9 to 15 (total duration: 14 days).
T½ of rosuvastatin | Blood samples for pharmacokinetic analyses will be taken at various time points from Day 1 to 7 and Day 9 to 15 (total duration: 14 days).

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idorsia Pharmaceuticals Ltd.
Locations (1):
- CEPHA s.r.o., Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Anliker-Ort M, Dingemanse J, Janu L, Kaufmann P. Effect of Daridorexant on the Pharmacokinetics of P-Glycoprotein Substrate Dabigatran Etexilate and Breast Cancer Resistance Protein Substrate Rosuvastatin in Healthy Subjects. Clin Drug Investig. 2023 Nov;43(11):827-837. doi: 10.1007/s40261-023-01310-6. Epub 2023 Oct 19. PMID 37858005